CLINICAL TRIAL: NCT00339664
Title: Pharmacological Analysis of Human Samples Collected in Clinical Trials Performed Outside of the Intramural National Cancer Institute
Brief Title: Analyses of Human Samples Collected in Clinical Trials
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903242; 03-C-N242; NCT00898196 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Leukemia, Myeloid; Neoplasm Metastasis; Leukemia, Lymphoid; Prostate Cancer
Keywords: Pharmacokinetics; Quantify; HPLC; LC/MS; Pharmacodynamics
MeSH Terms: conditions — Leukemia, Myeloid; Neoplasm Metastasis; Leukemia, Lymphoid; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- 1/ patients: Patients on approved clinical trials

SUMMARY:
Cancer patients in clinical trials donate various human samples (e.g., serum, plasma, blood, urine, feces, bile, saliva) for research purposes.

The purpose of this study is to conduct further analyses on these existing samples from clinical trials that are being performed outside of, but in collaboration with, the National Cancer Institute.

DETAILED DESCRIPTION:
Various human samples (e.g., serum, plasma, whole blood, erythrocytes, urine, feces, bile, and/or saliva) will be collected from cancer patients enrolled on approved clinical trials, in accordance with the local protocol. These trials are being conducted at outside institutions, in collaboration with the National Cancer Institute (NCI) and the samples will be sent to the NCI for pharmacological analysis, involving determination of parent drug and/or metabolite concentrations and subsequent pharmacokinetics and statistical data analysis. This study aims to further characterize the clinical pharmacokinetic behavior of select cancer therapeutics. Future collaborators will be added via the protocol amendment procedure.

ELIGIBILITY:
* INCLUSION CRITERIA:

Any patients entered on approved trials of cancer therapeutics or agents that are commonly administered to patients with cancer at institutions outside of the intramural NCI are eligible for inclusion, provided that they have consented to pharmacological analysis in the original consent form.

EXCLUSION CRITERIA:

None anticipated at this time.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patients entered on approved trials of cancer therapeutics or agents that are commonly administered to patients with cancer@@@
Sampling Method: Non-Probability Sample
Enrollment: 2579 (Actual)
Dates: Start 2003-07-02 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Drug and/or metabolite concentration | Ongoing
  To quantitate drug and/or metabolite concentrations in human blood samples

SECONDARY OUTCOMES:
Pharmacological behavior of agents | Ongoing
  To characterize the clinical pharmacological behavior of agents

CONTACTS AND LOCATIONS:
Overall Officials: William D Figg, Pharm.D., Principal Investigator — National Cancer Institute (NCI)
Locations (17):
- United States (15):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Case Western Reserve University, Cleveland, Ohio
  - University of Maryland at Amish Research Clinic, Lancaster, Lancaster, Pennsylvania
  - Abramson Cancer Center, University of Pennsylvania, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburg Cancer Institute, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - McGuire Veterans Administration Medical Center, Richmond, Virginia
  - Massey Cancer Center, Virginia Commonwealth University, Richmond, Virginia
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam